CLINICAL TRIAL: NCT05223803
Title: Phase 2 Randomized Total Eradication of Metastatic Lesions Following Definitive Radiation to the Prostate in de Novo oligometaStatic Prostate Cancer (TERPS) Trial
Brief Title: TERPS Trial for de Novo Oligometastic Prostate Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Responsible Party: Principal Investigator, Department of Radiation Oncology, Principal Investigator, University of Maryland, Baltimore
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HP-00098826
Record Dates: First submitted 2022-01-10; First posted 2022-02-04 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-11

CONDITIONS: Prostate Cancer; Oligometastatic Disease
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Best systemic therapy (BST) + primary prostate radiation (XRT) (Active Comparator)
  Interventions: Radiation: Prostate radiation (XRT); Drug: Systemic Therapy
- BST + XRT + SABR metastasis-directed therapy (MDT) (Active Comparator)
  Interventions: Radiation: Prostate radiation (XRT); Drug: Systemic Therapy; Radiation: Stereotactic ablative radiation therapy (SABR)

INTERVENTIONS:
Radiation: Prostate radiation (XRT) — Both arms will receive prostate radiation. Multiple treatment regimens are allowed per protocol.
Drug: Systemic Therapy — All systemic therapy is provided as best prescribed for patient per their medical oncologist.
Radiation: Stereotactic ablative radiation therapy (SABR) — SABR is delivered to those randomized to Arm 2.
  Arms: BST + XRT + SABR metastasis-directed therapy (MDT)

SUMMARY:
This research is being done to see if we can improve the outcome of prostate cancer patients who present with metastatic lesions at initial diagnosis.

DETAILED DESCRIPTION:
This study will compare the effects, good and/or bad, of using the standard of care treatment (systemic therapy + primary prostate radiation) compared to standard of care treatment plus stereotactic ablative radiation therapy (SABR) to metastatic lesions for prostate patients. The researchers are also trying to learn if the addition of SABR will affect recurrence rates. Presence of circulating tumor cells, gut bacteria, and quality of life will be assessed for both groups.

ELIGIBILITY:
Inclusion Criteria:

1. Patient must have at least one and up to three asymptomatic metastatic tumor(s) of the bone or soft tissue (with at least one bone metastasis) develop within the past 6-months that are seen on imaging. Up to five lesions are allowed on advanced functional imaging such as fluciclovine (Axumin), choline or PSMA PET-CT scan.

   1. CT or MRI scan within 6 months of enrollment
   2. Bone scan within 6 months of enrollment
   3. Fluciclovine (Axumin), choline, or PSMA PET-CT scan within 6 months of enrollment (PET-CT scan is reasonable for study entry imaging as an alternative to CT/MRI scan and bone scan)
2. Histologic confirmation of malignancy (primary or metastatic tumor).
3. Patient may have had prior systemic therapy and/or ADT associated with treatment within 9-months of enrollment.
4. PSA > 0.5 but <100.
5. Patient must be ≥ 18 years of age.
6. Patient must have a life expectancy ≥ 12 months.
7. Patient must have an ECOG performance status ≤ 2.
8. Patient must have the ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

1. Castration-resistant prostate cancer (CRPC).
2. Prior radiation therapy to an overlapping site of a target lesion that would preclude further radiation therapy
3. Spinal cord compression or impending spinal cord compression.
4. Suspected pulmonary and/or liver metastases (greater >10 mm in largest axis).
5. Patient receiving any other investigational agents.
6. Inability to receive any form of systemic therapy in the opinion of a treating medical oncologist .
7. Unable to lie flat during or tolerate PET/MRI, PET/CT or SABR.
8. No radiographical evidence of cranial metastasis.
9. Refusal to sign informed consent.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 122 (Estimated)
Dates: Start 2022-10-18 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2027-07-31 (Estimated)

PRIMARY OUTCOMES:
To determine the 2-year failure-free survival (FFS) of men who have oligometastatic prostate cancer with BST+XRT versus BST+XRT+SABR MDT. | 2 years
  Cross-over to the SABR MDT is allowed following failure.

SECONDARY OUTCOMES:
To determine the number of participants with toxicities related to SABR MDT in patients with de novo oligometastatic disease | 5 years
  Adverse events will be assessed at baseline, on treatment visit, and follow-up visit.
To determine local control at 12-months after SABR MDT in patients with de novo oligometastatic disease. | 1 year
To assess time to progression | 5 years
  Progression will be assessed for time to locoregional progression, time to distant progression, time to new metastasis, radiographic progression-free survival and duration of response after randomization to best systemic therapy (BST) and primary prostate radiation (XRT) versus BST, XRT and stereotactic ablative radiation therapy (SABR) metastasis-directed therapy (MDT).
Quality of life assessed through EPIC tool utilizing patient scores in each function group following completion of SABR MDT. | 5 years
  EPIC quality of life tool will be used to assess quality of life following treatment. This survey will be completed at baseline and during follow-up visits. Averages will be taken for each section in the survey (Urinary Function, Bowel Function, Sexual Function, and Hormonal function).

CONTACTS AND LOCATIONS:
Locations (9):
- United States (9):
  - UC San Diego Moores Cancer Center, La Jolla, California
  - Maryland Proton Treatment Center, Baltimore, Maryland
  - UMMC, Baltimore, Maryland
  - Upper Chesapeake Health, Bel Air, Maryland
  - Central Maryland Radiation Oncology, Columbia, Maryland
  - Baltimore Washington Medical Center, Glen Burnie, Maryland
  - Sidney Kimmel Cancer Center at Jefferson Health, Philadelphia, Pennsylvania
  - UPMC Hillman Cancer Center, Pittsburgh, Pennsylvania
  - Bon Secours Cancer Institute at St. Francis, Midlothian, Virginia

IPD SHARING:
Plan to Share IPD: No